CLINICAL TRIAL: NCT04049643
Title: Impact of Hearing Aid Intervention on Individuals With Cognitive Disorders
Brief Title: Hearing Aid and Individuals With Cognitive Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yu-Hsiang Wu (Other)
Collaborators: Vanderbilt University Medical Center (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor-Investigator, Yu-Hsiang Wu, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201907763; 3R01DC015997-02S1 (NIH)
Record Dates: First submitted 2019-08-06; First posted 2019-08-08 (Actual); Results first posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-03

CONDITIONS: Presbycusis, Bilateral; Alzheimer Disease 2 Due to Apoe4 Isoform; Mild Cognitive Impairment
Keywords: Presbycusis; Hearing aid; Alzheimer Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Presbycusis; Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Audiologist-Based (Active Comparator): In this group, the audiologist-based fitting will be used to provide hearing aids.
  Interventions: Device: Audiologist-based fitting
- Service-Only (Experimental): In this group, hearing aids that have minimum amplification will be fitted by audiologists.
  Interventions: Device: Service-only Fitting
- Device-Only (Experimental): In this group, hearing aids will be provided with minimum services from audiologists.
  Interventions: Device: Device-only fitting

INTERVENTIONS:
Device: Audiologist-based fitting — Hearing aids will be fitted by audiologists using established procedures.
  Arms: Audiologist-Based
Device: Service-only Fitting — This intervention group is designed to explore the contribution of amplification devices in hearing aid intervention, which consists of devices and services. In this intervention group, audiological services plus hearing aids that provide minimum amplification will be provided. Specifically, patient participants in this group will receive audiological services (e.g., counselling and education), except that the hearing aids will be set to provide no amplification other than what is needed to overcome any sounds that are dampened by the earpieces.
  Arms: Service-Only
Device: Device-only fitting — This intervention group is designed to explore the contribution of amplification devices in hearing aid intervention, which consists of devices and services. The patient participants in this intervention group will have minimum services regarding the pre-fitting, selection, and orientation of the hearing aids. The participants will have a hearing evaluation, including pure-tone audiometry. The audiologist will select the amplification characteristics and non-custom ear piece based on the audiogram. The audiologist will then briefly orient the participant on how to use the hearing aids and counsel on how to optimize their performance.
  Arms: Device-Only

SUMMARY:
This is a pilot study with the aim of evaluating the feasibility of the procedures of a future clinical trial that will help determine the impacts of hearing aid interventions on older patients with Alzheimer's Disease and related dementias (ADRD). In this pilot study individuals with mild or moderate cognitive impairment, as well as their caregivers, will be recruited. Participants will be randomly assigned to three intervention groups: Audiologist-Based Intervention, Service-Only Group, and Device-Only Group. Outcome data will be collected on the how hearing loss and hearing aid impact their lives and caregiver burden 6-week post hearing aid intervention.

DETAILED DESCRIPTION:
A disorder that often affect older adults is age-related hearing loss. It is estimated that about two-thirds of persons aged 70 years or older exhibit hearing problems. Left untreated, age-related hearing loss can affect an individual's ability to communicate and to interact with his/her environment and can contribute to psychological symptoms such depression, anxiety, isolation, paranoia, and possibly dementia.

Because (1) the neuropsychiatric symptoms associated with dementia could be exacerbated by poor communication resulting from hearing loss and (2) it has been widely accepted that hearing aids (HAs) are effective in improving communication function and reducing the psychosocial consequences associated with hearing loss for older adults without dementia, it seems reasonable to use HAs to treat the hearing loss of adults with Alzheimer's Disease and related dementias (ADRD). However, it has been argued that because the pathology of ADRD could involve central auditory pathways and nuclei, HAs-the devices that improve audibility at the peripheral level of the auditory system-may not be an effective management for ADRD. To date there is no high-quality evidence to support or negate the benefit of HA intervention on adults with dementia in reducing communication difficulty, dementia-related symptoms, and caregiver burdens. Therefore, the benefit of HA intervention on adults with ADRD remains unknown. Further, the best service model to provide HAs for older adults with ADRD is unknown. On one hand, it is likely that customized HAs fitted by audiologists using best practices could generate optimal outcomes. However, implementing the best-practice audiology services is challenging in this population. On the other hand, recent literature suggests that audiologists could fit low-cost, pre-programmed, non-customized amplification devices to adults with ADRD to reduce the cost of HA intervention, while yielding reasonable outcomes.To date there is no high-quality research rigorously examining the outcome, value, and candidacy of different HA service-delivery models for older adults with ADRD.

This is a pilot study with the aim of evaluating the feasibility of the procedures of a future clinical trial that will help determine the impacts of hearing aid interventions on older patients with ADRD. We expect that at least a total of 30 patients will complete the pilot study. The collected data will provide valuable information for us to formulate or revise the hypotheses, conduct power analysis, and finalize the research protocol for the future clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Montreal Cognitive Assessment (MoCA) score lower than 25 points
* Adult-onset mild-to-moderate sensorineural hearing loss

Exclusion Criteria:

* Non-native English speaker
* Prior hearing aid experience

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2024-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Hsiang Wu, PhD, Principal Investigator — University of Iowa
Locations (2):
- United States (2):
  - University of Iowa, Iowa City, Iowa
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
The proposed research will include data from participants with hearing loss recruited State of Iowa, State of Tennessee and surrounding areas. The final dataset will include self-reported demographic and behavioral data (e.g., questionnaire). Contact the principle investigator for data access.
Time Frame: The date will be available starting 6 months after publication of the main findings of the trial.
Access Criteria: Even though the final dataset will be stripped of identifiers prior to release for sharing, there remains the possibility of deductive disclosure of subjects with the survey data being collected. Thus, we will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate technologies; and (3) a commitment to destroying or returning the data after analyses are completed.

REFERENCES:
- [Background] Uhlmann RF, Larson EB, Rees TS, Koepsell TD, Duckert LG. Relationship of hearing impairment to dementia and cognitive dysfunction in older adults. JAMA. 1989 Apr 7;261(13):1916-9. PMID 2926927
- [Background] Palmer CV, Adams SW, Durrant JD, Bourgeois M, Rossi M. Managing hearing loss in a patient with Alzheimer disease. J Am Acad Audiol. 1998 Aug;9(4):275-84. PMID 9733237
- [Background] Palmer CV, Adams SW, Bourgeois M, Durrant J, Rossi M. Reduction in caregiver-identified problem behaviors in patients with Alzheimer disease post-hearing-aid fitting. J Speech Lang Hear Res. 1999 Apr;42(2):312-28. doi: 10.1044/jslhr.4202.312. PMID 10229449
- [Background] Mamo SK, Reed NS, Price C, Occhipinti D, Pletnikova A, Lin FR, Oh ES. Hearing Loss Treatment in Older Adults With Cognitive Impairment: A Systematic Review. J Speech Lang Hear Res. 2018 Oct 26;61(10):2589-2603. doi: 10.1044/2018_JSLHR-H-18-0077. PMID 30304320
- [Background] Loughrey DG, Kelly ME, Kelley GA, Brennan S, Lawlor BA. Association of Age-Related Hearing Loss With Cognitive Function, Cognitive Impairment, and Dementia: A Systematic Review and Meta-analysis. JAMA Otolaryngol Head Neck Surg. 2018 Feb 1;144(2):115-126. doi: 10.1001/jamaoto.2017.2513. PMID 29222544
- [Background] Livingston G, Sommerlad A, Orgeta V, Costafreda SG, Huntley J, Ames D, Ballard C, Banerjee S, Burns A, Cohen-Mansfield J, Cooper C, Fox N, Gitlin LN, Howard R, Kales HC, Larson EB, Ritchie K, Rockwood K, Sampson EL, Samus Q, Schneider LS, Selbaek G, Teri L, Mukadam N. Dementia prevention, intervention, and care. Lancet. 2017 Dec 16;390(10113):2673-2734. doi: 10.1016/S0140-6736(17)31363-6. Epub 2017 Jul 20. No abstract available. PMID 28735855
- [Background] Hopper T, Slaughter SE, Hodgetts B, Ostevik A, Ickert C. Hearing Loss and Cognitive-Communication Test Performance of Long-Term Care Residents With Dementia: Effects of Amplification. J Speech Lang Hear Res. 2016 Dec 1;59(6):1533-1542. doi: 10.1044/2016_JSLHR-H-15-0135. PMID 27973661
- [Background] Adrait A, Perrot X, Nguyen MF, Gueugnon M, Petitot C, Collet L, Roux A, Bonnefoy M; ADPHA study group. Do Hearing Aids Influence Behavioral and Psychological Symptoms of Dementia and Quality of Life in Hearing Impaired Alzheimer's Disease Patients and Their Caregivers? J Alzheimers Dis. 2017;58(1):109-121. doi: 10.3233/JAD-160792. PMID 28269769

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Audiologist-Based | Service-Only | Device-Only
Started | 9 | 3 | 5
Completed | 8 | 2 | 4
Not Completed | 1 | 1 | 1
Not completed — Lack of Efficacy | 1 | 1 | 0
Not completed — Health concern (unrelated to the intervention of the study) | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Audiologist-Based | Service-Only | Device-Only | Total
Number analyzed (Participants) | 8 | 2 | 4 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.4 (8.2) | 74 (1.4) | 60.5 (14.7) | 69 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 0 | 2
  Male | 6 | 2 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 2 | 4 | 14
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 8 | 2 | 4 | 14
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 2 | 4 | 14
Hearing loss (pure-tone average) [Mean (Standard Deviation); unit: dB HL] — Measure Description: Hearing loss measured using pure-tone audiometer. Pure-tone average is the mean of hearing threshold at 0.5, 1, and 2 kilohertz.
  dB HL | 36.8 (5.0) | 22.1 (4.1) | 21.9 (5.3) | 30.4 (8.9)

OUTCOME MEASURES:

1. Primary Outcome: Hearing Aid Benefit as Measured by the International Outcomes Inventory for Hearing Aids (IOI-HA)
Description: The IOI-HA is a questionnaire designed to assess the benefits of hearing aids from the user's perspective. The score ranges from 1 (less benefit) to 5 (more benefit).
Time Frame: 6 weeks after the first day participants started using hearing aids.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Audiologist-Based | Service-Only | Device-Only
Number analyzed (Participants) | 8 | 2 | 4
score on a scale | 3.9 (0.6) | 3.4 (0.3) | 3.7 (0.6)

2. Primary Outcome: Change of Daily Activity as Measured by the Lawton Instrumental Activities of Daily Living Scale (IADL)
Description: The IADL was developed to assess independent living skills, such as feeding, dressing, and food preparation. The score ranges from 0 (low function) to 8 (high function). Participants complete this measure pre-intervention and at 6 weeks post-intervention. The change in scores between pre- and post-intervention are reported, with score changes ranging from +8 (indicating a benefit from hearing aids) to -8 (indicating a detrimental effect of hearing aids).
Time Frame: Immediately before hearing aid use and 6 weeks after the first day of hearing aid use
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Audiologist-Based | Service-Only | Device-Only
Number analyzed (Participants) | 8 | 2 | 4
score on a scale | 1 (5) | 0 (0) | 0 (0)

3. Primary Outcome: Change of Caregiver Burden as Measured by the "Zarit Burden Interview" (ZBI)
Description: Caregiver burden will be measured using the ZBI, which is a 22-item questionnaire. The ZBI measures self-reported burden in terms of the degree (from 'never' to 'almost always') to which the caregiver experiences physical, psychological, emotional, social and financial problems as a result of their care-giving role. The score ranges from 0 (little or no burden) to 88 (severe burden). This measure is completed pre-intervention and at 6 weeks post-intervention. The change in scores between pre- and post-intervention are reported, with score changes ranging from -88 (indicating a benefit from hearing aids) to +88 (indicating a detrimental effect of hearing aids).
Time Frame: Immediately before hearing aid use and 6 weeks after the first day of hearing aid use
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Audiologist-Based | Service-Only | Device-Only
Number analyzed (Participants) | 8 | 2 | 4
score on a scale | -2.6 (5.5) | -7 (2.8) | -1 (7.9)

4. Secondary Outcome: Change of Hearing Handicap Measured by Hearing Handicap Inventory for the Elderly (HHIE) or Hearing Handicap Inventory for Adults (HHIA)
Description: The HHIE and HHIA are questionnaires designed to measure perceived hearing handicap. For subjects order and younger 65 years old, the HHIE and HHIA will be used, respectively. The score ranges from 0 (no handicap) to 100 (more handicap) (i.e., lower scores mean less handicap). Participants will complete this questionnaire pre-intervention and at 6 weeks post-intervention. The change in scores between pre- and post-intervention are reported, with score changes ranging from -100 (indicating a benefit from hearing aids) to +100 (indicating a detrimental effect of hearing aids).
Time Frame: Immediately before hearing aid use and 6 weeks after the first day of hearing aid use
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Audiologist-Based | Service-Only | Device-Only
Number analyzed (Participants) | 6 | 2 | 4
score on a scale | -36 (20.1) | -14 (11.3) | -17.5 (21.7)

5. Secondary Outcome: Change of Quality of Life as Measured by the Alzheimer's Disease-Related Quality of Life (ADRQL)
Description: The ADRQL was developed to assess health related quality of life in people with Alzheimer's disease using assessments from family caregivers or professional staff. The score ranges from 0 (worst situation) to 100 (best situation). Participants complete this measure pre-intervention and at 6 weeks post-intervention. The change in scores between pre- and post-intervention are reported, with score changes ranging from +100 (indicating a benefit from hearing aids) to -100 (indicating a detrimental effect of hearing aids).
Time Frame: Immediately before hearing aid use and 6 weeks after the first day of hearing aid use
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Audiologist-Based | Service-Only | Device-Only
Number analyzed (Participants) | 8 | 2 | 4
score on a scale | 5.0 (8.3) | 13.8 (30) | 1.25 (3.9)

6. Secondary Outcome: Change of Depression as Measured Using the Geriatric Depression Scale (GDS)
Description: The GDS a self-report measure of depression in older adults. The short form of the GDS has 15 items. The score ranges from 0 (no depression) to 15 (more depression) Participants complete this measure pre-intervention and at 6 weeks post-intervention. The change in scores between pre- and post-intervention are reported, with score changes ranging from -15 (indicating a benefit from hearing aids) to +15 (indicating a detrimental effect of hearing aids).
Time Frame: Immediately before hearing aid use and 6 weeks after the first day of hearing aid use
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Audiologist-Based | Service-Only | Device-Only
Number analyzed (Participants) | 7 | 2 | 3
score on a scale | -0.85 (2.4) | 0.5 (0.7) | -0.33 (0.57)

ADVERSE EVENTS:
Time Frame: Adverse events are monitored for each subject during their participation in the study, which averaged 7 weeks from the time the participants entered the study.
Arm/Group | Audiologist-Based | Service-Only | Device-Only
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/2 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/2 | 0/4
Other Adverse Events (participants affected / at risk) | 0/8 | 0/2 | 0/4

LIMITATIONS AND CAVEATS:
This study faced challenges in recruiting subjects for the Service-Only and Device-Only groups. Since blinding was not feasible, some potential participants chose not to provide consent after learning their group assignment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-10-01): https://cdn.clinicaltrials.gov/large-docs/43/NCT04049643/Prot_SAP_002.pdf
  • Informed Consent Form (2022-01-24): https://cdn.clinicaltrials.gov/large-docs/43/NCT04049643/ICF_000.pdf